CLINICAL TRIAL: NCT05903625
Title: Effect of Lysine and Phosphorous in Double Fortified Bread on Glycemic Index (GI) of White Bread and Postprandial Glycemia
Brief Title: Effect of Lysine and Phosphorus Fortification on Glycemic Index and Postprandial Glycemia in Double Fortified Bread
Acronym: LP-DFB-GI-PG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Mahnoor, MPhil Scholar, UVAS, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Double Salt UVAS
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hyperglycemia; Glucose Metabolism Disorders; Metabolic Disease; Glycemic Index
Keywords: Glycemic Index; Postprandial Glycemia; Lysine; Phosphorus; White bread; Glycemic Control
MeSH Terms: conditions — Hyperglycemia; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Lysine

STUDY DESIGN:
Intervention Model Description: This clinical trial utilizes a cross-over design, administering multiple interventions to the same group of participants. The interventions include standard white bread, lysine-fortified bread, phosphorous-fortified bread, and a combination of lysine and phosphorous-fortified bread. Each participant receives these interventions in a specific sequence, with a washout period between each one to eliminate residual effects. This design allows for within-subject comparisons and minimizes individual variability. By examining the effects on glycemic index and postprandial glycemia, the cross-over design provides comprehensive insights. It enhances efficiency, statistical power, and enables the exploration of treatment interactions. Overall, this cross-over design allows for a thorough investigation of the impact of these interventions on glycemic index and postprandial glycemia in the study's participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group - Standard White Bread (Experimental): This arm serves as the control group in the clinical trial, providing a baseline comparison for the intervention arms. Participants in this arm consume standard white bread
  Interventions: Dietary Supplement: Control Group - Standard White Bread
- Lysine Group - Lysine-Fortified Bread (Experimental): This arm investigates the effect of lysine-fortified bread on glycemic response. Participants in this arm consume bread fortified with lysine, an essential amino acid.
  Interventions: Dietary Supplement: Lysine Group - Lysine-Fortified Bread
- Phosphorus Group - Phosphorus-Fortified Bread (Experimental): This arm explores the impact of phosphorus-fortified bread on glycemic response. Participants in this arm consume bread fortified with phosphorus, an essential mineral.
  Interventions: Dietary Supplement: Phosphorus Group - Phosphorus-Fortified Bread
- Lysine and Phosphorus Group - Double Fortified Bread (Experimental): This arm examines the combined effect of lysine and phosphorus in double fortified bread on glycemic response. Participants in this arm consume bread fortified with both lysine and phosphorus.
  Interventions: Dietary Supplement: Lysine and Phosphorus Group - Double Fortified Bread

INTERVENTIONS:
Dietary Supplement: Control Group - Standard White Bread — Participants consume commercially available standard white bread, serving as the control intervention.
  Arms: Control Group - Standard White Bread
Dietary Supplement: Lysine Group - Lysine-Fortified Bread — Participants consume bread fortified with lysine, an essential amino acid, in a specified dosage, frequency, and duration.
  Arms: Lysine Group - Lysine-Fortified Bread
Dietary Supplement: Phosphorus Group - Phosphorus-Fortified Bread — Participants consume bread fortified with phosphorus, an essential mineral, in a specified dosage, frequency, and duration
  Arms: Phosphorus Group - Phosphorus-Fortified Bread
Dietary Supplement: Lysine and Phosphorus Group - Double Fortified Bread — Double Fortified Bread: Participants consume bread fortified with both lysine and phosphorus in specified dosages, frequencies, and durations.
  Arms: Lysine and Phosphorus Group - Double Fortified Bread

SUMMARY:
The goal of this clinical trial is to investigate the effect of lysine and phosphorous on the glycemic index (GI) of white bread and postprandial glycemia. The main questions it aims to answer are:

* Can double fortification with lysine and phosphorous lower the glycemic index (GI) of bread?
* Does double fortification with lysine and phosphorous improve postprandial glycemia?

Participants in the study will be assigned to the control group, where they will consume regular white bread, then to the experimental group, where they will consume double fortified bread with lysine and phosphorous. The glycemic response of the bread samples will be measured by monitoring blood glucose levels in healthy participants after consuming the bread. The glycemic index will also be calculated based on the area under the curve (AUC) of the test food compared to a standard. The collected data will be analyzed using statistical methods such as paired sample t-tests and one-way ANOVA.

The expected outcomes of the study are that lysine and phosphorous will reduce the glycemic index of white bread and also decrease the postprandial blood glucose spike. This research aims to provide valuable insights into fortifying bread to improve its health impact, particularly for individuals with diabetes or at risk of developing diabetes

DETAILED DESCRIPTION:
This study aims to investigate the effect of lysine and phosphorous in double fortified bread on the glycemic index (GI) of white bread and postprandial glycemia. The research will be conducted through a human trial involving 16 participants. The study protocol includes the objectives, design, methods, scientific background, and statistical considerations.

The objective of the study is to evaluate the impact of lysine and phosphorous fortification on the glycemic response to bread consumption. The study will employ a interventional study design with four intervention groups. The participants will be assigned into Group 1 (simple white bread), Group 2 (lysine fortified bread), Group 3 (phosphorous fortified bread), and Group 4 (lysine and phosphorous fortified bread).

To ensure accurate measurements, the study will involve multiple readings at different time intervals. Blood glucose levels will be measured at 15 minutes, 30 minutes, 45 minutes, 90 and 120 minutes after consuming the bread. Each experiment will be conducted for a single group on a specific date. Each experiment will be repeated with a three-day gap between each repetition. This schedule ensures that each group receives the intervention on separate days and allows for sufficient time between experiments to minimize any carryover effects or potential confounding factors. Baseline fasting blood glucose levels will also be assessed before consuming the test foods.

The primary outcomes of the study are the glycemic index (GI) and postprandial glycemia. The glycemic index will be calculated through incremental area under the curve (iAUC) of the test food to that of standard food. The iAUC values will be compared between the intervention groups to assess the effects of lysine and phosphorous fortification on glycemic response.

The statistical analysis plan will include descriptive statistics to summarize participant characteristics and baseline variables. Statistical tests such as analysis of variance (ANOVA) or non-parametric equivalent tests will be used to compare the intervention groups.

The time frame for the study will focus on the immediate post-meal period, typically within 2 hour, to evaluate the acute effects of the bread interventions on blood glucose levels. The study protocol takes into account ethical considerations, participant recruitment, informed consent, data collection procedures, and data analysis methods.

The scientific background of the study includes a review of existing literature on the effects of lysine and phosphorous on glycemic response. It provides a rationale for investigating the specific research question and highlights the potential implications of the study findings.

Overall, the study protocol outlines a rigorous and systematic approach to investigate the effect of lysine and phosphorous fortification on the glycemic index and postprandial glycemia of white bread. The detailed description ensures clarity and transparency in the research methodology, allowing researchers, participants, and data users to understand the objectives, design, methods, and statistical considerations of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are appropriate if they are in the age range between 18 and 35 years.
* Subjects should be within normal range of BMI 18.5 to 24.5 kg per meter square.
* Efforts will be made to age and gender match subjects

Exclusion Criteria:

* Subjects with diabetes, cardiovascular, cerebrovascular, pulmonary, hepatic, renal, endocrinological (PTH), or any significant medical disease will be excluded.
* Pregnant and lactating women.
* Subjects on regular use of any medication and supplements.
* Subjects that have any type of food allergy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Measure 1 - Postprandial Glycemia | 120 minutes of post-meal consumption
  Postprandial glycemia will be assessed at specific time intervals following the consumption of the test foods. The blood glucose levels will be measured using standardized methods, such as finger prick blood glucose testing using glucometer. The postprandial glycemia metric provides valuable information about the short-term effects of the different bread interventions on blood glucose regulation and response
Measure 2- Glycemic Index (GI) of the white bread | up to 12 weeks
  Glycemic Index is determined by measuring the rise in blood glucose levels over a specific time period after consuming a fixed amount of the test food, compared to a reference food (usually glucose or white bread). The GI value is expressed as a percentage or a numerical scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mah Noor, MPhil, Principal Investigator — University of Veterinary and Animal Sciences, Lahore
Locations (1):
- University of Veterinary and Animal Sciences, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang L, Li X. [Level of serum phosphorus and adult type 2 diabetes mellitus]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2016 May;41(5):502-6. doi: 10.11817/j.issn.1672-7347.2016.05.009. Chinese. PMID 27269925
- [Background] Jozi F, Kheiripour N, Taheri MA, Ardjmand A, Ghavipanjeh G, Nasehi Z, Shahaboddin ME. L-Lysine Ameliorates Diabetic Nephropathy in Rats with Streptozotocin-Induced Diabetes Mellitus. Biomed Res Int. 2022 Sep 12;2022:4547312. doi: 10.1155/2022/4547312. eCollection 2022. PMID 36132073
- [Background] Bahmani F, Bathaie SZ, Aldavood SJ, Ghahghaei A. Prevention of alpha-crystallin glycation and aggregation using l-lysine results in the inhibition of in vitro catalase heat-induced-aggregation and suppression of cataract formation in the diabetic rat. Int J Biol Macromol. 2019 Jul 1;132:1200-1207. doi: 10.1016/j.ijbiomac.2019.04.037. Epub 2019 Apr 6. PMID 30965074
- [Background] Khattab M, Abi-Rashed C, Ghattas H, Hlais S, Obeid O. Phosphorus ingestion improves oral glucose tolerance of healthy male subjects: a crossover experiment. Nutr J. 2015 Oct 29;14:112. doi: 10.1186/s12937-015-0101-5. PMID 26514124
- [Background] Kalogeropoulou D, LaFave L, Schweim K, Gannon MC, Nuttall FQ. Lysine ingestion markedly attenuates the glucose response to ingested glucose without a change in insulin response. Am J Clin Nutr. 2009 Aug;90(2):314-20. doi: 10.3945/ajcn.2008.27381. Epub 2009 Jun 24. PMID 19553295
- [Background] Jordi J, Herzog B, Lutz TA, Verrey F. Novel antidiabetic nutrients identified by in vivo screening for gastric secretion and emptying regulation in rats. Am J Physiol Regul Integr Comp Physiol. 2014 Oct 1;307(7):R869-78. doi: 10.1152/ajpregu.00273.2014. Epub 2014 Aug 6. PMID 25100072
- See also: This interventional clinical trial aims to assess the effects of fortifying white flour with lysine and/or phosphorus on postprandial glycemia and energy expenditure. — http://www.clinicaltrials.gov/ct2/show/NCT03836495